CLINICAL TRIAL: NCT02331225
Title: Endothelial Mircroparticles as a Biomarker of Pulmonary Hypertension in Systemic Sclerosis
Brief Title: Endothelial Microparticles in Systemic Sclerosis Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: University of South Alabama (Other)
Responsible Party: Principal Investigator, Matthew Lammi, Assistant Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: 8772
Record Dates: First submitted 2014-12-18; First posted 2015-01-06 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Systemic Sclerosis; Pulmonary Hypertension; Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Systemic sclerosis, no pulmonary hypertension: This group will be systemic sclerosis patients without pulmonary hypertension
  Interventions: Other: No intervention given
- Systemic sclerosis/pulmonary hypertension: This group will be systemic sclerosis patients with pulmonary hypertension
  Interventions: Other: No intervention given
- Healthy controls: These will be healthy age- and sex-matched controls
  Interventions: Other: No intervention given

INTERVENTIONS:
Other: No intervention given — There is no intervention for this study

SUMMARY:
Systemic sclerosis (SSc, also known as scleroderma) is a disease characterized by fibrosis of the skin and organs, inflammation, and an abnormal endothelial cell lining inside of vessels. A common and deadly complication of SSc is pulmonary hypertension (PH), which is an abnormal elevation in the blood pressure within the lung blood vessels. Early identification and treatment of PH is important in SSc, and no clinical factors can predict which patients will develop PH with acceptable accuracy. A potential marker of PH in SSc is the presence of increased amounts of endothelial microparticles (EMPs), which are substances circulating in the blood that were released from damaged vessel wall endothelial lining. A main goal of this study is to investigate if there is a difference in EMP levels between SSc patients with and without PH. The investigators will also use human endothelial cells in a lab environment to test whether these EMPs isolated from SSc patients are actually causing damage to the vessel lining. Lastly, the investigators will investigate the potential benefit of a medication used after transplant, mycophenolate mofetil (MMF). This will be done by causing damage to isolated human endothelial cells and treating them with MMF. The main goal of this portion of our study is to see if EMP levels are reduced when cells are treated with MMF. Overall, the investigators anticipate the following outcomes of this study: 1) use EMP levels to differentiation patients with SSc who have PH from those without PH, 2) use EMPs to understand how endothelial damage occurs in SSc, and 3) use EMPs to help us develop new treatments for patients with vascular diseases.

ELIGIBILITY:
For systemic sclerosis subjects:

Inclusion Criteria:

* Age >18 years
* Meet American College of Rheumatology criteria for systemic sclerosis

Exclusion Criteria:

* Chronic kidney disease (estimated creatinine clearance <50mL/min)
* Uncontrolled hypertension (diastolic blood pressure>120mmHg)
* Acute coronary syndrome within the past 6 months
* Chronic obstructive pulmonary disease
* Diabetes mellitus
* Hemolytic anemia
* Active tobacco abuse

For healthy control subjects:

Inclusion Criteria:

* Age>18 years
* Age- and sex-matched to SSc patients

Exclusion criteria:

* Coronary artery disease
* Uncontrolled hypertension (diastolic blood pressure>120mmHg)
* Chronic obstructive pulmonary disease
* Chronic kidney disease
* Diabetes mellitus
* Hemolytic anemia
* Active tobacco abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be 3 groups: systemic sclerosis subjects with pulmonary hypertension, systemic sclerosis subjects without pulmonary hypertension, and healthy age- and sex-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Plasma VE-cadherin + endothelial microparticle levels | Baseline
  endothelial microparticles are expressed as microparticles per microliter of plasma. This is a cross-sectional analysis, so the measurements will be performed once, on study visit 1

SECONDARY OUTCOMES:
Plasma PECAM+ endothelial microparticles | Baseline
  endothelial microparticles are expressed as microparticles per microliter of plasma. This is a cross-sectional analysis, so the measurements will be performed once, on study visit 1
Plasma E-selectin + endothelial microparticles | Baseline
  endothelial microparticles are expressed as microparticles per microliter of plasma. This is a cross-sectional analysis, so the measurements will be performed once, on study visit 1

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Health Sciences Center, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Tual-Chalot S, Guibert C, Muller B, Savineau JP, Andriantsitohaina R, Martinez MC. Circulating microparticles from pulmonary hypertensive rats induce endothelial dysfunction. Am J Respir Crit Care Med. 2010 Jul 15;182(2):261-8. doi: 10.1164/rccm.200909-1347OC. Epub 2010 Mar 25. PMID 20339146
- [Background] Guiducci S, Distler JH, Jungel A, Huscher D, Huber LC, Michel BA, Gay RE, Pisetsky DS, Gay S, Matucci-Cerinic M, Distler O. The relationship between plasma microparticles and disease manifestations in patients with systemic sclerosis. Arthritis Rheum. 2008 Sep;58(9):2845-53. doi: 10.1002/art.23735. PMID 18759303
- [Background] Iversen LV, Ostergaard O, Ullman S, Nielsen CT, Halberg P, Karlsmark T, Heegaard NH, Jacobsen S. Circulating microparticles and plasma levels of soluble E- and P-selectins in patients with systemic sclerosis. Scand J Rheumatol. 2013;42(6):473-82. doi: 10.3109/03009742.2013.796403. Epub 2013 Sep 9. PMID 24016306
- [Background] Amabile N, Heiss C, Real WM, Minasi P, McGlothlin D, Rame EJ, Grossman W, De Marco T, Yeghiazarians Y. Circulating endothelial microparticle levels predict hemodynamic severity of pulmonary hypertension. Am J Respir Crit Care Med. 2008 Jun 1;177(11):1268-75. doi: 10.1164/rccm.200710-1458OC. Epub 2008 Feb 28. PMID 18310479
- [Background] Amabile N, Heiss C, Chang V, Angeli FS, Damon L, Rame EJ, McGlothlin D, Grossman W, De Marco T, Yeghiazarians Y. Increased CD62e(+) endothelial microparticle levels predict poor outcome in pulmonary hypertension patients. J Heart Lung Transplant. 2009 Oct;28(10):1081-6. doi: 10.1016/j.healun.2009.06.005. PMID 19782291
- [Derived] Lammi MR, Saketkoo LA, Okpechi SC, Ghonim MA, Wyczechowska D, Bauer N, Pyakurel K, Saito S, deBoisblanc BP, Boulares AH. Microparticles in systemic sclerosis: Potential pro-inflammatory mediators and pulmonary hypertension biomarkers. Respirology. 2019 Jul;24(7):675-683. doi: 10.1111/resp.13500. Epub 2019 Feb 12. PMID 30747487